CLINICAL TRIAL: NCT06415838
Title: Behavioral Activation for the Prevention and Treatment of Depression in Older Adults in a Municipal Context: a Randomized Controlled Trial
Brief Title: Behavioral Activation for the Prevention and Treatment of Depression in Older Adults in a Municipal Context
Acronym: DePrevent
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sormland County Council, Sweden (Other)
Collaborators: Eskilstuna municipality (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DePrevent
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Depression; Depressive Symptoms
Keywords: Behavioral activation; Behavior therapy; Psychological treatment; Older adults; Geriatric
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brief Behavioral Activation plus Care as Usual (Experimental): Five-session Brief Behavioral Activation intervention. Sessions 1 - 4 are completed once a week, and session 5 is a booster-session completed four weeks after session 4.
  Interventions: Behavioral: Brief Behavioral Activation; Other: Care as Usual
- Care as Usual (Active Comparator): Care as usual as provided by primary care and/or municipal care.
  Interventions: Other: Care as Usual

INTERVENTIONS:
Behavioral: Brief Behavioral Activation — A five-session brief behavioral activation treatment delivered face-to-face in the participants' home.
  Session outline:
  Session 1: Psychoeducation about depression; treatment rationale for Behavioral Activation (BA); rationale and instructions for activity log
  Session 2: Discussion of life goals and values; planning of activities aligned with life goals and values for coming week
  Session 3: Troubleshooting any problems carrying out activities; planning activities aligned with life goals and values for coming week.
  Session 4: Troubleshooting any problems carrying out activities; planning activities aligned with life goals and values for the coming week; instructing the participant to independently continue to plan activities for the coming month.
  Session 5: Troubleshooting any problems carrying out activities; reviewing treatment; stressing the importance of continuing to engage in activities aligned with life goals and values; creating a maintenance plan.
  Arms: Brief Behavioral Activation plus Care as Usual
Other: Care as Usual — Care as Usual provided by primary care and/or municipal care.

SUMMARY:
The goal of this randomized clinical trial is to investigate if a brief psychological treatment called Behavioral Activation (BA) works to prevent and treat depression in older adults in a municipal context in Sweden. It will also learn about the patients' and therapists' experiences of the BA-treatment.

The main questions it aims to answer are if the BA-treatment has an effect on the short and long term on:

* Depressive symptoms
* Anxiety symptoms
* Self-rated activation
* Functional ability
* Loneliness
* Self efficacy
* Mental wellbeing
* Quality of life
* Need for community care services

All participants will continue their care as usual (CAU), and half of the participants will be randomized to receive a five-session BA-treatment spread over two months as an add-on to CAU. All participants will answer a questionnaire in the beginning of the study, after two months, and after 3-, 6- and 12 months.

DETAILED DESCRIPTION:
One third of the Swedish population aged 70 years and above report depressive symptoms, and between 5 - 15% have a major depressive disorder. Depression in older adults reduces quality of life and functional ability, and is associated with an increased risk for morbidity and mortality. Psychological treatment is considered a first-line treatment for depression, but is currently only offered to about 3% of older adults with depression in Sweden. A majority of older adults suffering from depression in Sweden are likely not to be identified and diagnosed, and thereby not treated for their depression. Furthermore, many older adults receive municipal care, and psychological treatment is currently not available in this context.

The goal of this randomized clinical trial is to investigate if a brief psychological treatment called Behavioral Activation (BA) works to prevent and treat depression in older adults in a municipal context in Sweden. It will also learn about the patients' and therapists' experiences of the BA-treatment. The therapists in the trial are social workers working in Eskilstuna municipality in Sweden.

All participants will continue their care as usual (CAU), and half of the participants will be randomized to receive a five-session BA-treatment spread over two months as an add-on to CAU. The BA-treatment will be delivered in the participants' home. All participants will answer a questionnaire in the beginning of the study, after two months, and after 3-, 6- and 12 months.

The main questions that the trial aims to answer are if the BA-treatment has an effect on the short and long term on:

* Depressive symptoms
* Anxiety symptoms
* Self-rated activation
* Functional ability
* Loneliness
* Self efficacy
* Mental wellbeing
* Quality of life
* Need for community care services

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* 5 points or above on the Geriatric Depression Scale 15, GDS-15
* Fluent in written and spoken Swedish
* Consents to participate in the trial

Exclusion Criteria:

* Not able to use the patient materials due to visual impairment
* Not able to communicate with therapist due to hearing impairment
* Diagnosis of major neurocognitive disorder
* Below 25 points on the Mini Mental State Examination, MMSE
* Elevated suicide risk
* Current substance- or alcohol use disorder
* Previous or current psychotic disorder
* Previous or current bipolar disorder
* Ongoing psychological treatment/pscyhotherapy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale, MADRS-S | Baseline; post-intervention or equivalent for control group 9 weeks after baseline; 3-, 6- and 12 months post-intervention or equivalent for control group
  Depressive symptoms will be measured with the Montgomery-Åsberg Depression Rating Self-rating Scale (MADRS-S). The MADRS-S is a nine-item questionnaire designed to measure depression severity during the past two weeks. The total score ranges from 0-54, with higher scores indicating higher depression severity.

SECONDARY OUTCOMES:
Geriatric Depression Scale 15, GDS-15 | Baseline; post-intervention or equivalent for control group 9 weeks after baseline; 3-, 6- and 12 months post-intervention or equivalent for control group
  Depressive symptoms and depression diagnoses will also be measured using the Geriatric Depression Rating Scale 15-item short form (GDS-15), a 15-item questionnaire used to identify depression in older individuals with scores ranging from 0-15, with higher scores indicating higher depression severity.
Geriatric Anxiety Scale 10, GAS-10 | Baseline; post-intervention or equivalent for control group 9 weeks after baseline; 3-, 6- and 12 months post-intervention or equivalent for control group
  Anxiety symptoms will be measured with the Geriatric Anxiety Scale - 10 item version (GAS-10), with a score ranging from 0 - 30, with higher scores indicating higher levels of anxiety.
WHO disability assessment schedule 12-item, WHODAS-12 | Baseline; post-intervention or equivalent for control group 9 weeks after baseline; 3-, 6- and 12 months post-intervention or equivalent for control group
  Functional impairment will be assessed with the WHO Disability Assessment Schedule 12-item (WHODAS-12), a self-rating scale with 12 items ranging from 0 - 48, with higher scores indicating more functional impairment.
Behavioral activation for depression scale - short form, BADS-SF | Baseline; post-intervention or equivalent for control group 9 weeks after baseline; 3-, 6- and 12 months post-intervention or equivalent for control group
  Self-rated avoidance and activation will be measured using the Behavioral Activation for Depression Scale - Short Form (BADS-SF), a 9-item scale with scores ranging from 0 - 54, with higher scores indicating a higher degree of activation and lower degree of avoidance.
UCLA Loneliness Scale version 3, UCLA-LS 3 | Baseline; post-intervention or equivalent for control group 9 weeks after baseline; 3-, 6- and 12 months post-intervention or equivalent for control group
  Subjective feelings of loneliness and social isolation will be measured using the UCLA Loneliness Scale version 3 (UCLA-LS 3), a 20-item scale with scores ranging from 20 - 80 points, with higher scores indicating higher loneliness.
The New General Self-Efficacy Scale, S-GSE | Baseline; post-intervention or equivalent for control group 9 weeks after baseline; 3-, 6- and 12 months post-intervention or equivalent for control group
  New General Self-Efficacy Scale (S-GSE) is an 10-item measure with scores ranging between 10 - 40 points, that assesses how much people believe they can achieve their goals, despite difficulties. Higher scores indicate higher levels of self-efficacy.
EuroQol-5 Dimensions-5 Level Scale, EQ-5D-5L | Baseline; post-intervention or equivalent for control group 9 weeks after baseline; 3-, 6- and 12 months post-intervention or equivalent for control group
  Health related quality of life and estimation of quality-adjusted life years (QALY) for health economic evaluations will be measured using the EuroQol-5 Dimensions-5 Level Scale (EQ-5D-5L), a 5-item scale ranging between 1 - 5 per item, measuring health status with regards to mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The Eq-5D-5L also has an overall health scale where the rater selects a number between 1-100 to describe the condition of their health, with higher scores indicating better overall health.
Short Warwick-Edinburgh Mental Wellbeing Scale, SWEMWBS | Baseline; post-intervention or equivalent for control group 9 weeks after baseline; 3-, 6- and 12 months post-intervention or equivalent for control group
  Self-rated mental wellbeing will be measured with the Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS), a 7-item scale with scores ranging from 7 - 35, with higher scores indicating higher positive mental wellbeing.
Need for municipal care service | Baseline; post-intervention or equivalent for control group 9 weeks after baseline; 3-, 6- and 12 months post-intervention or equivalent for control group
  Need for municipal care service will be measured by recording types of services and number of hours granted by the municipality for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Johnny Pellas, PhD, Principal Investigator — Research and Development Sormland
Locations (1):
- Eskilstuna kommun, Eskilstuna, Sörmland, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol and statistical analysis plan to be shared/published before data collection has ended.